CLINICAL TRIAL: NCT04897373
Title: The Effects of an Active Older Adult Program at the Dan Abraham Healthy Living Center on Health and Well-being
Brief Title: Active Older Adult Program on Health and Well-being
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Nathan K. LeBrasseur, Principal Investigator, Mayo Clinic
Other Study IDs: 18-001769
Record Dates: First submitted 2021-05-17; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Older Adult

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood-derived plasma and CD3+ T-cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine whether a structured 12-week program designed for older adults will improve physical function and, in parallel, circulating biomarkers of aging

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 55 years or older.
* Membership at the DAHLC.
* New to AOA (Active Older Adult) Program and commitment to full participation in the twelve-week program.
* Must be able to get down and off the floor with little assistance.

Exclusion Criteria:

* Inability to provide informed consent.
* Previous participation in the AOA Program at the DAHLC.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population consists of The Dan Abraham Healthy Living Center (DAHLC) members 60 years of age and older who plan to participate in the Active Older Adult Program.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
Change in repeated chair rise time | Baseline to end of study, approximately 14 weeks
  Chair stand test where participants will perform a chair rise movement for five repetitions. The series of 5 repetitions will be timed and measured in seconds.
Change in plasma protein levels reflective of biological age | Baseline, week 12
  Blood samples will be obtained at baseline and at 12 weeks. The concentration of target proteins (pg/mL) in the plasma will be measured and compared between baseline and week 12.
Change in expression of senescence-related genes in blood cells | Baseline, week 12
  Blood samples will be obtained at baseline and at 12 weeks. The expression of senescence-related genes (arbitrary units) will be measured in immune cells isolated from whole blood and compared between baseline and week 12.

SECONDARY OUTCOMES:
Change in Self-reported Physical Function | Baseline, week 12
  Measured using the Physical Component Scale (PCS) from the 12-Item short form general health survey (SF-12).
Change in Performance-based Physical Function | Baseline, week 12
  Measured using the timed up-and-go test (seconds to complete).
Change in Mental Function | Baseline, week 12
  Measured using the Mental Component Scale (MCS) from the 12-Item short form general health survey (SF-12)
Change in self-assessment of well-being | Baseline, week 12
  Measured using a linear analogue self-assessment scale of well-being from 0 ("as bad as it can be") to 10 ("as good as it can be") of mental, physical, emotional, and spiritual well-being, level of social activity, and overall quality of life during the past week

CONTACTS AND LOCATIONS:
Overall Officials: Nathan LeBrasseur, PhD, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials